CLINICAL TRIAL: NCT02201784
Title: A Comparative Study Between Levobupivacaine 0.5% and Ropivacaine 0.75% in Patients Undergoing Spinal Anaesthesia for Lower Limb Orthopaedic Surgery.
Brief Title: Spinal Anaesthesia With Levobupivacaine 0.5% and Ropivacaine 0.75% for Lower Limb Orthopaedic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aligarh Muslim University (Other)
Responsible Party: Principal Investigator, MANAZIR ATHAR, Doctor, Aligarh Muslim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jnmch2012
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Lower Limb Surgery
Keywords: Subarachnoid block; intrathecal; spinal anesthesia; isobaric; levobupivacaine; ropivacaine
MeSH Terms: interventions — Levobupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine 0.5% (Active Comparator): intrathecal administration of 15 mg of Levobupivacaine 0.5%
  Interventions: Drug: Levobupivacaine
- Ropivacaine 0.75% (Active Comparator): intrathecal administration of 22.5 mg of Ropivacaine 0.75%
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Comparison of Equipotent doses
  Other Names: Chirocaine
  Arms: Levobupivacaine 0.5%
Drug: Ropivacaine — Comparison of equipotent doses
  Other Names: Naropin
  Arms: Ropivacaine 0.75%

SUMMARY:
The purpose of this study is to compare the effects of two intrathecally administered drugs:0.5% levobupivacaine and0.75%Ropivacaine in spinal anesthesia

DETAILED DESCRIPTION:
Bupivacaine is a highly cardiotoxic drug and also produces prolonged motor blockade.The newer drugs levobupivacaine and ropivacaine being comparatively less cardio and neurotoxic are preferred now a days.So, we conducted this prospective, randomized double blind study with an aim of comparing the efficacy and characteristics of these drugs.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) class I & II patients of either sex
2. Age between 18-60 years

Exclusion Criteria:

1. Patient's refusal.
2. Patients who have contraindications to spinal anaesthesia / Local anaesthetic drugs.
3. Patients having h/o diabetes, neurological and musculoskeletal diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manazir Athar, M.D, Principal Investigator — Jawaharlal Nehru Medical College, AMU,Aligarh, India; Syed Moied Ahmed, PhD, M.D, Study Director — Jawaharlal Nehru Medical College, AMU, Aligarh, India; Masood H Siddiqi, M.S, Study Director — Jawaharlal Nehru Medical College, AMU, Aligarh, India
Locations (1):
- Jawaharlal Nehru medical college, AMU, Aligarh, Uttar Pradesh, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: jawaharlal nehru medical college and hospital
Pre-assignment Details: Patients who met any of the exclusion criteria or those who did not gave consent were excluded.
Period: Overall Study
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75%
Started | 30 | 30
Completed | 28 | 30
Not Completed | 2 | 0
Not completed — Failure to achieve adequate block | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75% | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (17) | 35 (16) | 37 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 24 | 23 | 47
Region of Enrollment [Number; unit: participants]
  India | 30 | 30 | 60
Weight [Mean (Standard Deviation); unit: kg] | 53.83 (9.44) | 57.17 (6.65) | 55.5 (8.27)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia
Description: Defined as time for first analgesic request by the patient
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75%
Number analyzed (Participants) | 28 | 30
minutes | 309.83 (36.45) | 249.50 (22.83)

2. Secondary Outcome: Onset of Sensory Block at T10
Description: level of sensory block was assessed every 5 minutes till the loss of sensation to pinprick, using 22-guage hypodermic needle with 2mm protrusion through guard. Assessments continued at 30 min intervals following the completion of surgery until normal sensation returned.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75%
Number analyzed (Participants) | 28 | 30
minutes | 13.50 (4.94) | 7.33 (2.54)

3. Secondary Outcome: Median Maximum Level of Sensory Blockade
Description: as for outcome 2
Time Frame: 8 hours
Reporting Status: Not Posted

4. Secondary Outcome: Time to Maximum Cephalic Spread of Sensory Block
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75%
Number analyzed (Participants) | 28 | 30
minutes | 20.33 (5.31) | 13.17 (3.02)

5. Secondary Outcome: Onset of Motor Block to Bromage3
Description: Motor block in the lower limbs was graded according to the modified Bromage scale (Grade 0 = No motor block, Grade 1 = Inability to raise extended leg, able to move knees and feet, Grade 2 = Inability to raise extended leg and move knee, able to move feet, Grade 3 = Complete motor block of the lower limbs). Thereafter, It was performed every 5 minutes till the attainment of MB grade 3 followed by every 30 minutes until complete recovery (MB grade0).
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75%
Number analyzed (Participants) | 28 | 30
minutes | 12.17 (4.09) | 7.83 (2.84)

6. Secondary Outcome: Duration of Motor Block
Description: Time when the Bromage score will be back to zero
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75%
Number analyzed (Participants) | 28 | 30
minutes | 290.50 (34.67) | 222.50 (23.00)

7. Other Pre Specified Outcome: Pulse Rate, Mean Arterial Pressure, SpO2
Description: Intragroup and intergroup variation compared
Time Frame: 8 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Levobupivacaine 0.5% | Ropivacaine 0.75%
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/30 | 13/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levobupivacaine 0.5% (N=30) | Ropivacaine 0.75% (N=30)
Nausea (Gastrointestinal disorders) | 4 | 2
Bradycardia (Cardiac disorders) | 2 | 2 — Heart rate was recorded before induction, every 3 min till 15 minutes, then, every 15 min until discharge from the recovery room.Bradycardia was defined as HR<50 beat/min
Shivering (General disorders) | 3 | 5
Hypotension (Cardiac disorders) | 7 | 10 — Arterial blood pressure was recorded before induction, every 3 min till 15 minutes, then, every 15 min until discharge from the recovery room. Hypotension was defined as systolic BP < 90 mm Hg

LIMITATIONS AND CAVEATS:
Exact baricity was not known as Specific gravity was not measured; Quality of anaesthesia was not assessed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No